CLINICAL TRIAL: NCT05017233
Title: Spectral CT Clinical Trial Protocol
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigational product had been released in NMPA, Sponsor decided to terminate the study aligned with investigator
Sponsor: Philips (China) Investment CO., LTD (Industry)
Collaborators: Shanghai Changzheng Hospital (Other); Ruijin Hospital (Other); West China Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PD_CT_Hawk_2021_11258
Record Dates: First submitted 2021-08-10; First posted 2021-08-23 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: CT Scanning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Experimental group, all volunteer will be scanned. (Experimental): All participation accept Spectral CT scanning; No group;
  Interventions: Device: Spectral CT

INTERVENTIONS:
Device: Spectral CT — Using Spectral CT to scan Breast

SUMMARY:
The purpose of this study was to evaluate the expected effectiveness, ease of operation, stability, and safety of Spectral CT

DETAILED DESCRIPTION:
Under the premise of protecting subjects and ensuring the scientific nature of this study, Spectral CT was evaluated for its effectiveness, convenience, stability and safety under normal conditions by collecting clinical cases.

ELIGIBILITY:
Inclusion Criteria:

* Recruit volunteers (ages 18 to 75);
* Negative pregnancy tests in women of childbearing age;
* Participants who agree to participate in this clinical trial and sign the informed consent;
* Enhanced scans require laboratory tests to confirm normal renal function.

Exclusion Criteria:

* Persons who do not have full capacity for civil conduct;
* Lactating women;
* People who are not suitable for enhanced scanning with iodine contrast agent;
* Patients whom the investigator considers inappropriate to participate in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Excellent and good rate of clinical imaging (score≥3） | through study completion, an average of 1 year
  Rated items 5 points Excellent image quality for diagnostic purposes, very satisfactory 4 points good image quality, can be used for diagnosis, satisfactory 3 points Image quality defects, do not affect the diagnosis, general 2. Unsatisfactory image quality, affecting diagnosis Poor image quality, undiagnosable, unsatisfactory

SECONDARY OUTCOMES:
Common functions assessment | through study completion, an average of 1 year
  Common function evaluation items inclduing:The exposure function; Bed body moving; Microphone intercom function; Image post-processing function; Data storage management. With Satisfied, normal, Not Satisfied
Convenience evaluation assessment | through study completion, an average of 1 year
  Convenience function evaluation items inclduing:Laser positioning lamp Breathing navigation Control buttons The clinical interface friendliness of postprocessing software The post-processing software is convenient for clinical use and operation. With Satisfied, normal, Not Satisfied
Machine function and stability assessment | through study completion, an average of 1 year
  Machine function and stability evaluation items inclduing:workflow Image display and transmission Failed to start system Unexpected system shutdown Abnormal termination during the scan Unable to expose during scan. With Satisfied, normal, Not Satisfied
Adverse events and serious adverse events | through study completion, an average of 1 year
  Adverse events and serious adverse events during the test were collected to evaluate the safety of the product.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyuan Liu, Director, Principal Investigator — Shanghai Changzheng Hospital; Fuhua Yan, Director, Principal Investigator — Ruijin Hospital; Bin Song, Director, Principal Investigator — West China Hospital
Locations (3):
- China (3):
  - West China Hospital, Chengdu, Sichuan
  - Ruijin Hospital, Shanghai
  - Shanghai Changzheng Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: No